CLINICAL TRIAL: NCT04491240
Title: The Protocol of Evaluation of Safety and Efficiency of Method of Exosome Inhalation in SARS-CoV-2 Associated Two-Sided Pneumonia
Brief Title: Evaluation of Safety and Efficiency of Method of Exosome Inhalation in SARS-CoV-2 Associated Pneumonia.
Acronym: COVID-19EXO
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: State-Financed Health Facility "Samara Regional Medical Center Dinasty" (Other)
Collaborators: Samara State Medical University (Other); Samara Regional Clinical Hospital V.D. Seredavin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: COVID-19 EXO
Record Dates: First submitted 2020-07-27; First posted 2020-07-29 (Actual); Results first posted 2020-11-04 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-10

CONDITIONS: Covid19; SARS-CoV-2 PNEUMONIA; COVID-19
Keywords: Covid-19; SARS-CoV-2; exosomes; MSC
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: The trial has three groups, each with 10 subjects (n=30). All eligible study subjects will be randomized, double-blinded, to either the two treatment groups or placebo group.
Who Masked: Participant, Care Provider
Masking Description: Two main groups will be provided with exosomes in a specially provided solution, the third group (control) will receive the same solution without exosomes. Due to exosomes are nanoparticles and requires special methods and devices to be detected the hospital staff and patients have no way to check which group receives exosomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EXO-1 (Experimental): Participants (n=10) in this group will receive standard therapy and exosomes of the first type.
  Interventions: Drug: EXO 1 inhalation
- EXO-2 (Experimental): Participants (n=10) in this group will receive standard therapy and exosomes of the second type.
  Interventions: Drug: EXO 2 inhalation
- Placebo (Placebo Comparator): Participants (n=10) in this group will receive standard therapy and inhalation placebo solution.
  Interventions: Drug: Placebo inhalation

INTERVENTIONS:
Drug: EXO 1 inhalation — Twice a day during 10 days inhalation of 3 ml special solution contained 0.5-2x10^10 of nanoparticles (exosomes) of the first type.
  Arms: EXO-1
Drug: EXO 2 inhalation — Twice a day during 10 days inhalation of 3 ml special solution contained 0.5-2x10^10 of nanoparticles (exosomes) of the second type.
  Arms: EXO-2
Drug: Placebo inhalation — Twice a day during 10 days inhalation of 3 ml special solution free of nanoparticles (exosomes).
  Arms: Placebo

SUMMARY:
Coronavirus is an acute viral disease with prevailing upper respiratory tract infections caused by the RNA-containing virus of the genus Betacoronavirus of the Coronaviridae family. Most patients with severe COVID-19 develop pneumonia in the first week of the disease. As the infection progresses, the infiltration increases, and the affected areas increases. Excessive and uncontrolled immune system response with rapidly developing fatal cytokine storm plays the main role in the pathogenesis of acute respiratory distress syndrome (ARDS) due to SARS-CoV-2 infection.

According to available data, exosomes can regulate inflammation and regenerative processes due to the change in the concentration of anti-inflammatory cytokines and switch the immune cell to regenerative secretome. Inhalation of exosomes may reduce inflammation and damage to the lung tissue and stimulate the regenerative processes.

This protocol has been developed based on the literature, information about the ongoing tests NCT04276987 (A Pilot Clinical Study on Inhalation of Mesenchymal Stem Cells Exosomes Treating Severe Novel Coronavirus Pneumonia) and NCT04384445 (Organicell Flow for Patients With COVID-19), Patent No 271036826 of 2019. "A method for obtaining and concentrating microRNA-containing exosomal multi-potent mesenchymal-stromal cells for use in cosmetic and pharmaceutical products to stimulate regenerative processes and slow down aging.

DETAILED DESCRIPTION:
COVID-19 is an infectious disease caused by the most recently discovered coronavirus. This new virus and disease were unknown before the outbreak began in Wuhan, China, in December 2019. COVID-19 is now a pandemic affecting many countries worldwide. Globally, as of 1:09 pm CEST, 27 July 2020, there have been 16 096 741 confirmed cases of COVID-19, including 646 384 deaths, reported to WHO.

The main and rapidly achievable target of SARS-CoV-2 is lung type II alveolar cells (AT2), which determines the development of diffuse alveolar damage. In the pathogenesis of ARDS due to COVID-19, the main role is played by an over-response of the immune system with rapidly developing severe life-threatening cytokine release syndrome (cytokine storm). Cytokine release syndrome threatens the emergence and progression of ARDS. The key components of the pathogenesis of ARDS also include disruption of cell cytotoxicity mechanisms, excessive activation of cytotoxic lymphocytes and macrophages with a massive release of proinflammatory cytokines (FNO-α, IL-1, IL-2, IL-6, IL-8, IL-10), granulocytic colony-stimulating factor, monocytic chemoattractive protein 1), and inflammatory markers (CRP, serum ferritin), infiltration of internal organs and tissues by activated T-lymphocytes and macrophages, resulting in a hyperinflammatory reaction. Such severe lesions can lead to death or severe lung damage, including long rehabilitation after discharge.

Experimental studies have demonstrated that mesenchymal stem cells (MSCs) may significantly reduce lung inflammation and pathological impairment resulting from different types of lung injury. Many researchers connect the anti-inflammatory effect of MSC with their secretome which includes MSC derived exosomes. It is highly likely that MSC exosomes have the same therapeutic effect on inoculation pneumonia as MSCs themselves. Moreover, exosomes show a strong effect of regenerative stimulation on different wounds so the regenerative effect can be extended on patients with COVID-19 pneumonia.

The purpose of this protocol is to explore the safety and efficiency of aerosol inhalation of the exosomes in the treatment of severe patients hospitalized with novel coronavirus pneumonia (NCP).

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand the study objectives and risks and provide signed and dated informed consent;
* Confirmed COVID-19 infection (by PCR or antibody test);
* Pneumonia requiring hospitalization, and oxygen saturation of <94% indoors or a need for auxiliary oxygen. The confirmed volume of lung damage by CT: not less than 30% and not more than 80%;
* ability to proceed with inhalation by self;

Exclusion Criteria:

* Severe respiratory failure at the time of screening due to COVID-19 pneumonia;
* Known to undergo medical resuscitation for 14 days before randomization;
* Any serious medical condition or deviation of the clinical laboratory parameter that, in the opinion of the researcher, prevents safe participation and completion of the study by the participant Confirmed uncontrolled active bacterial, fungal, viral or other infection (other than SARS-CoV-2).
* According to the researcher, the progression to death is inevitable and will occur within the next 24 hours, regardless of the therapy.
* The life expectancy of fewer than 28 days, taking into account a medical condition already existing that cannot be corrected, e.g. participants with the following conditions or suspicions: polyorganic insufficiency, poorly controlled neoplasms, terminal stage heart disease, cardiopulmonary cardiac arrest that required cardiopulmonary resuscitation, or electrical activity not accompanied by a pulse, or asystole within the last 30 days, terminal stage liver disease, terminal stage liver disease, or liver disease;
* Pregnancy or breastfeeding;
* Liver function failure (Class C for Child-Pugh), detected within 24 hours at screening (local laboratory);
* Absolute neutrophil count (ANC) <500 cells/µL at screening (local laboratory);
* Platelet count <50000 cells/µL at screening (based on laboratory data);
* Creatinine level ≥ 1.5 from the upper limit;
* Uncontrolled or untreated arrhythmia with clinical manifestations, myocardial infarction within the last 6 weeks or congestive heart failure (NYHA Degrees 3 or 4);
* Respiratory failure in the last 6 months or home use of oxygen in severe chronic respiratory disease (COPD);
* Quadriplegia;
* Primary immunodeficiency, tuberculosis, progressive multifocal leukoencephalopathy, aspergillosis or other invasive mold/fungal infection in anamnesis, or internal or bone marrow transplantation for 6 months before randomization;
* Known infection with hepatitis B or C viruses requiring therapy;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Centre Dinasty, Samara, Russia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | EXO-1 | EXO-2 | Placebo
Started | 10 | 10 | 10
Completed | 10 | 10 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EXO-1 | EXO-2 | Placebo | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 10 | 30
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 47.9 [29 to 62] | 52.5 [39 to 60] | 53.3 [38 to 64] | 51.23 [29 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 5 | 19
  Male | 4 | 2 | 5 | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Russia | 10 | 10 | 10 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Non-serious and Serious Adverse Events During Trial
Description: Safety assessment such as adverse events will be registered. Adverse events will be monitored during all trial
Time Frame: 30 days after clinic discharge
Measure: Count of Participants; unit: Participants
Arm/Group | EXO-1 | EXO-2 | Placebo
Number analyzed (Participants) | 10 | 10 | 10
Participants
  Number of participants with serious adverse events during trial | 0 | 0 | 0
  Number of participants with non-serious adverse events during trial | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Non-serious and Serious Adverse During Inhalation Procedure
Description: Safety assessments such as adverse events during the inhalation procedures will be registered.
Time Frame: after each inhalation during 10 days
Measure: Count of Participants; unit: Participants
Arm/Group | EXO-1 | EXO-2 | Placebo
Number analyzed (Participants) | 10 | 10 | 10
Participants
  Temperature increase | 0 | 0 | 0
  Bronchospasm | 0 | 0 | 0
  allergic reaction in the form of swelling Quincke, rash, seizures, etc. | 0 | 0 | 0
  Other | 0 | 0 | 0

3. Secondary Outcome: Time to Clinical Recovery (TTCR)
Description: Measure and compare time to clinical recovery compared to placebo. Time to clinical recovery calculated by the number of days the patient has hospitalized.
Time Frame: from first inhalation until discharge from the clinic, up to 30 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | EXO-1 | EXO-2 | Placebo
Number analyzed (Participants) | 10 | 10 | 10
days | 13.8 (1.55) | 14.8 (2.35) | 14.1 (1.37)

4. Secondary Outcome: SpO2 Concentration
Description: The concentration of SpO2 by Pulse oximetry device during procedures in the groups. The measure was done before and after each inhalation (total 4 measures per day). The intraday SpO2 data of all patients in groups was calculated as Median with Inter-Quartile Range and presented in the table by days.
Time Frame: 10 days during inhalation
Measure: Median (Inter-Quartile Range); unit: O2 concentration in percent
Arm/Group | EXO-1 | EXO-2 | Placebo
Number analyzed (Participants) | 10 | 10 | 10
O2 concentration in percent
  Day 1 | 93.8 [93.5 to 94] | 94.5 [93.6 to 94.9] | 94 [94 to 94.9]
  Day 2 | 94.8 [94 to 95] | 95.3 [94.1 to 95.9] | 96 [95.6 to 96]
  Day 3 | 95.3 [95 to 95.5] | 95.5 [94.6 to 95.9] | 96 [95.1 to 96.4]
  Day 4 | 95.5 [95.1 to 95.9] | 96 [95.6 to 96.9] | 96.5 [96 to 96.9]
  Day 5 | 96 [95.3 to 96.4] | 96.5 [95.6 to 96.9] | 97.3 [96.6 to 97.5]
  Day 6 | 96 [96 to 96.9] | 97 [96.3 to 97] | 97 [97 to 97.5]
  Day 7 | 96.8 [96.5 to 97.5] | 97.5 [97 to 97.5] | 97.5 [97 to 97.9]
  Day 8 | 97.3 [97 to 98] | 97.3 [97 to 97.9] | 98.3 [97.1 to 98.9]
  Day 9 | 97.3 [97 to 98] | 97.8 [97 to 99] | 98.5 [98.1 to 98.9]
  Day 10 | 97.8 [97.1 to 98.8] | 98.5 [97.6 to 99] | 98.8 [98 to 99]

5. Secondary Outcome: C-reactive Protein
Description: Blood biochemistry C reactive protein level in serum.
Time Frame: At the begining of inhalation (day 1) and on next day of last inhalation (day 11)
Measure: Mean (Full Range); unit: mg/L
Arm/Group | EXO-1 | EXO-2 | Placebo
Number analyzed (Participants) | 10 | 10 | 10
mg/L
  Day 1 | 78.3 [4.3 to 299] | 75.4 [5.7 to 137] | 61.5 [11.6 to 147]
  Day 11 | 5.04 [0.5 to 12.5] | 5.83 [0.4 to 32.1] | 8.29 [0.4 to 41.1]
Statistical Analysis 1: Comparison: EXO-1; The study results were statistically processed using STATA version 9.0, Statistica for Windows version 6.0. Changes from the beginning of inhalation and after were compared using the T-test for depended group criterion, data between the main group and the control group were compared using the non-parametric method, box-plot. The data in the table presented as a Mean with full range (min-max). The difference calculated as Mean difference with 95% confidence interval and Standard Deviation (SD); Test type: Superiority; p = 0.020875, t-test, 2 sided; Mean Difference (Net) = 73.29000, 95% CI 2-sided [13.97687 to 132.6031], Standard Deviation 82.91404
Statistical Analysis 2: Comparison: EXO-2; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.000953, t-test, 2 sided; Mean Difference (Net) = 69.56000, 95% CI 2-sided [36.88502 to 102.2350], Standard Deviation 45.67648
Statistical Analysis 3: Comparison: Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.002233, t-test, 2 sided; Mean Difference (Net) = 53.21000, 95% CI 2-sided [24.69923 to 81.72077], Standard Deviation 39.85531

6. Secondary Outcome: Lactic Acid Dehydrogenase (LDH)
Description: Lactic Acid Dehydrogenase (LDH) level in serum
Time Frame: At the beginning of inhalation (day 1) and on next day of last inhalation (day 11)
Measure: Mean (Full Range); unit: U/L
Arm/Group | EXO-1 | EXO-2 | Placebo
Number analyzed (Participants) | 10 | 10 | 10
U/L
  at Day 1 | 773 [383 to 1285] | 732 [380 to 1867] | 669 [333 to 1260]
  at Day 11 | 441 [280 to 740] | 365 [30.4 to 648] | 430 [306 to 686]
Statistical Analysis 1: Comparison: EXO-1; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.008948, t-test, 2 sided; Mean Difference (Net) = 331.5200, 95% CI 2-sided [105.5938 to 557.4462], Standard Deviation 315.8230
Statistical Analysis 2: Comparison: EXO-2; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.020921, t-test, 2 sided; Mean Difference (Net) = 366.6300, 95% CI 2-sided [69.77651 to 663.4835], Standard Deviation 414.9726
Statistical Analysis 3: Comparison: Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.004873, t-test, 2 sided; Mean Difference (Net) = 239.2000, 95% CI 2-sided [93.20037 to 385.1996], Standard Deviation 204.0934

ADVERSE EVENTS:
Time Frame: During medical procedures and 1-month post-discharge from the clinic.
Description: Collection of information on unwanted reactions to inhalation after each inhalation, e.g. 1) temperature increase, 2) allergic reaction in the form of Quincke's disease, rash, seizures, etc.; 3) bronchospasm for inhalation.
Arm/Group | EXO-1 | EXO-2 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EXO-1 (N=10) | EXO-2 (N=10) | Placebo (N=10)
Temperature increase (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) — Increase in body temperature after each inhalation.
Allergic reactions (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) — Allergic reactions in the form of Quincke's disease, rash, seizures were assessed after each inhalation.
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) — bronchospasm for inhalation after the procedure were assessed after inhalation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-06): https://cdn.clinicaltrials.gov/large-docs/40/NCT04491240/Prot_SAP_000.pdf